CLINICAL TRIAL: NCT00757601
Title: A Single Dose Clinical Trial to Study the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of MK1006.
Brief Title: A Study to Test the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MK1006 (MK-1006-002)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1006-002; 2008_549
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- 15 mg MK1006/Placebo/45 mg MK1006/60 mg MK1006/Placebo (Fed) (Experimental): Participants received 15 mg MK1006 in Period 1, followed by placebo to MK1006 in Period 2, followed by 45 mg MK1006 in Period 3, followed by 60 mg MK1006 in Period 4, followed by placebo to MK1006 taken with food (Fed state) in Period 5.
  Interventions: Drug: MK1006; Drug: Placebo
- Placebo/30mg MK1006/45mg MK1006/60mg MK1006/30mg MK1006 (Fed) (Experimental): Participants received placebo to MK1006 in Period 1, followed by 30 mg MK1006 in Period 2, followed by 45 mg MK1006 in Period 3, followed by 60 mg MK1006 in Period 4, followed by 30 mg MK1006 taken with food (Fed state) in Period 5.
  Interventions: Drug: MK1006; Drug: Placebo
- 15mg MK1006/30mg MK1006/Placebo/60mg MK1006/30mg MK1006 (Fed) (Experimental): Participants received 15 mg MK1006 in Period 1, followed by 30 mg MK1006 in Period 2, followed by placebo to MK1006 in Period 3, followed by 60 mg MK1006 in Period 4, followed by 30 mg MK1006 taken with food (Fed state) in Period 5.
  Interventions: Drug: MK1006; Drug: Placebo
- 15mg MK1006/30mg MK1006/45mg MK1006/Placebo/30mg MK1006 (Fed) (Experimental): Participants received 15 mg MK1006 in Period 1, followed by 30 mg MK1006 in Period 2, followed by 45 mg MK1006 in Period 3, followed by placebo to MK1006 in Period 4, followed by 30 mg MK1006 taken with food (Fed state) in Period 5.
  Interventions: Drug: MK1006; Drug: Placebo
- 60mg MK1006 / Placebo / 100mg MK1006 / 120mg MK1006 / Placebo (Experimental): Participants received 60 mg MK1006 in Period 1, followed by placebo to MK1006 in Period 2, followed by 100 mg MK1006 in Period 3, followed by 120 mg MK1006 in Period 4, followed by placebo to MK1006 in Period 5.
  Interventions: Drug: MK1006; Drug: Placebo
- Placebo/ 80mg MK1006/ 100mg MK1006/ 120mg MK1006/ 140mg MK1006 (Experimental): Participants received placebo to MK1006 in Period 1, followed by 80 mg MK1006 in Period 2, followed by 100 mg MK1006 in Period 3, followed by 120 mg MK1006 in Period 4, followed by 140 mg MK1006 in Period 5
  Interventions: Drug: MK1006; Drug: Placebo
- 60mg MK1006/ 80mg MK1006/ Placebo/ 120mg MK1006/ 140mg MK1006 (Experimental): Participants received 60 mg MK1006 in Period 1, followed by 80 mg MK1006 in Period 2, followed by placebo to MK1006 in Period 3, followed by 120 mg MK1006 in Period 4, followed by 140 mg MK1006 in Period 5.
  Interventions: Drug: MK1006; Drug: Placebo
- 60mg MK1006/ 80mg MK1006/ 100mg MK1006/ Placebo/ 140mg MK1006 (Experimental): Participants received 60 mg MK1006 in Period 1, followed by 80 mg MK1006 in Period 2, followed by 100 mg MK1006 in Period 3, followed by placebo to MK1006 in Period 4, followed by 140 mg MK1006 in Period 5.
  Interventions: Drug: MK1006; Drug: Placebo
- 140mg MK1006 / Placebo / 200mg MK1006 / 230mg MK1006 / Placebo (Experimental): Participants received 140 mg MK1006 in Period 1, followed by placebo to MK1006 in Period 2, followed by 200 mg MK1006 in Period 3, followed by 230 mg MK1006 in Period 4, followed by placebo to MK1006 in Period 5.
  Interventions: Drug: MK1006; Drug: Placebo
- Placebo/170mg MK1006/ 200mg MK1006/ 230mg MK1006/ 260mg MK1006 (Experimental): Participants received placebo to MK1006 in Period 1, followed by 170 mg MK1006 in Period 2, followed by 200 mg MK1006 in Period 3, followed by 230 mg MK1006 in Period 4, followed by 260 mg MK1006 in Period 5.
  Interventions: Drug: MK1006; Drug: Placebo
- 140mg MK1006/170mg MK1006/ Placebo/ 230mg MK1006/ 260mg MK1006 (Experimental): Participants received 140 mg MK1006 in Period 1, followed by 170 mg MK1006 in Period 2, followed by placebo to MK1006 in Period 3, followed by 230 mg MK1006 in Period 4, followed by 260 mg MK1006 in Period 5
  Interventions: Drug: MK1006; Drug: Placebo
- 140mg MK1006/170mg MK1006/ 200mg MK1006/ Placebo/ 260mg MK1006 (Experimental): Participants received 140 mg MK1006 in Period 1, followed by 170 mg MK1006 in Period 2, followed by 200 mg MK1006 in Period 3, followed by placebo to MK1006 in Period 4, followed by 260 mg MK1006 in Period 5.
  Interventions: Drug: MK1006; Drug: Placebo

INTERVENTIONS:
Drug: MK1006 — MK1006 capsules: 1 mg, 10 mg, and 20 mg.
  Panel A: MK1006 capsules in five doses beginning at 15 mg and rising to 60 mg
  Panel B: MK1006 capsules in five doses beginning at 60 mg and rising to 140 mg.
  Panel C: MK1006 capsules in five doses beginning at 140 mg and rising to 260 mg.
  There will a 7-day interval between each dose
Drug: Placebo — Placebo capsule to match MK1006 1, 10, and 20 mg.
  Panel A: Placebo to MK1006 capsules in five doses beginning at 15 mg and rising to 60 mg
  Panel B: Placebo to MK1006 capsules in five doses beginning at 60 mg and rising to 140 mg.
  Panel C: Placebo to MK1006 capsules in 5 doses beginning at 140 mg and rising to 260 mg.
  There will a 7-day interval between each dose

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of single doses of MK1006

ELIGIBILITY:
Inclusion Criteria:

* Participant is between 18 and 55 years of age. Participants up to 65 years of age may be enrolled in Panels B and C
* Female participants must be postmenopausal or otherwise unable to have children
* Participant has a body mass index (BMI) less than or equal to 42 kg/m^2 at the screening visit
* Participant has type 2 diabetes and is being treated with either diet and exercise or a single oral anti-hyperglycemic medication. For Panels B and C, participant may be treated with combination oral anti-hyperglycemic medications
* Participant is willing to follow the American Heart Association (AHA) diet and exercise program throughout the study
* Participant is a nonsmoker or has not used nicotine-containing products for 6 months prior to study start

Exclusion Criteria:

* Participant has a history of stroke, seizures, or other neurological disorders
* Participant has a recent history of eye infection or other inflammatory eye conditions
* Participant has glaucoma or is blind
* Participant has had eye surgery within 6 months of study start (Lasik is permitted)
* Participant has type 1 diabetes
* Participant cannot stop taking any of their current prescription or non-prescription medications during the study
* Participant consumes more than 3 alcoholic beverages per day
* Participant consumes more than 6 caffeinated beverages per day
* Participant has had major surgery or has donated blood within 4 weeks of study start
* Participant has multiple and/or severe allergies to drugs or food

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- 15mg MK1006/Placebo/45mg MK1006/60mg MK1006/Placebo (Fed): Participants received 15 mg MK1006 in Period 1, followed by placebo to MK1006 in Period 2, followed by 45 mg MK1006 in Period 3, followed by 60 mg MK1006 in Period 4, followed by placebo to MK1006 taken with food (Fed state) in Period 5.
- Placebo/80mg MK1006/100mg MK1006/120mg MK1006/140mg MK1006: Participants received placebo to MK1006 in Period 1, followed by 80 mg MK1006 in Period 2, followed by 100 mg MK1006 in Period 3, followed by 120 mg MK1006 in Period 4, followed by 140 mg MK1006 in Period 5.
- 60mg MK1006/80mg MK1006/Placebo/120mg MK1006/140mg MK1006: Participants received 60 mg MK1006 in Period 1, followed by 80 mg MK1006 in Period 2, followed by placebo to MK1006 in Period 3, followed by 120 mg MK1006 in Period 4, followed by 140 mg MK1006 in Period 5.
- 60 mg MK1006/80 mg MK1006/100 mg MK1006/Placebo/140 mg MK1006: Participants received 60 mg MK1006 in Period 1, followed by 80 mg MK1006 in Period 2, followed by 100 mg MK1006 in Period 3, followed by placebo to MK1006 in Period 4, followed by 140 mg MK1006 in Period 5.
- Placebo/170mg MK1006/200mg MK1006/230mg MK1006/260mg MK1006: Participants received placebo to MK1006 in Period 1, followed by 170 mg MK1006 in Period 2, followed by 200 mg MK1006 in Period 3, followed by 230 mg MK1006 in Period 4, followed by 260 mg MK1006 in Period 5.
- 140mg MK1006/170mg MK1006/Placebo/230mg MK1006/260mg MK1006: Participants received 140 mg MK1006 in Period 1, followed by 170 mg MK1006 in Period 2, followed by placebo to MK1006 in Period 3, followed by 230 mg MK1006 in Period 4, followed by 260 mg MK1006 in Period 5.
- 140mg MK1006/170mg MK1006/200mg MK1006/Placebo/260mg MK1006: Participants received 140 mg MK1006 in Period 1, followed by 170 mg MK1006 in Period 2, followed by 200 mg MK1006 in Period 3, followed by placebo to MK1006 in Period 4, followed by 260 mg MK1006 in Period 5.
Period: Period 1
Arm/Group | 15mg MK1006/Placebo/45mg MK1006/60mg MK1006/Placebo (Fed) | Placebo/30mg MK1006/45mg MK1006/60mg MK1006/30mg MK1006 (Fed) | 15mg MK1006/30mg MK1006/Placebo/60mg MK1006/30mg MK1006 (Fed) | 15mg MK1006/30mg MK1006/45mg MK1006/Placebo/30mg MK1006 (Fed) | 60mg MK1006 / Placebo / 100mg MK1006 / 120mg MK1006 / Placebo | Placebo/80mg MK1006/100mg MK1006/120mg MK1006/140mg MK1006 | 60mg MK1006/80mg MK1006/Placebo/120mg MK1006/140mg MK1006 | 60 mg MK1006/80 mg MK1006/100 mg MK1006/Placebo/140 mg MK1006 | 140mg MK1006 / Placebo / 200mg MK1006 / 230mg MK1006 / Placebo | Placebo/170mg MK1006/200mg MK1006/230mg MK1006/260mg MK1006 | 140mg MK1006/170mg MK1006/Placebo/230mg MK1006/260mg MK1006 | 140mg MK1006/170mg MK1006/200mg MK1006/Placebo/260mg MK1006
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | 15mg MK1006/Placebo/45mg MK1006/60mg MK1006/Placebo (Fed) | Placebo/30mg MK1006/45mg MK1006/60mg MK1006/30mg MK1006 (Fed) | 15mg MK1006/30mg MK1006/Placebo/60mg MK1006/30mg MK1006 (Fed) | 15mg MK1006/30mg MK1006/45mg MK1006/Placebo/30mg MK1006 (Fed) | 60mg MK1006 / Placebo / 100mg MK1006 / 120mg MK1006 / Placebo | Placebo/80mg MK1006/100mg MK1006/120mg MK1006/140mg MK1006 | 60mg MK1006/80mg MK1006/Placebo/120mg MK1006/140mg MK1006 | 60 mg MK1006/80 mg MK1006/100 mg MK1006/Placebo/140 mg MK1006 | 140mg MK1006 / Placebo / 200mg MK1006 / 230mg MK1006 / Placebo | Placebo/170mg MK1006/200mg MK1006/230mg MK1006/260mg MK1006 | 140mg MK1006/170mg MK1006/Placebo/230mg MK1006/260mg MK1006 | 140mg MK1006/170mg MK1006/200mg MK1006/Placebo/260mg MK1006
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 (One participant discontinued the study after Period 2 and was replaced by another participant.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 3
Arm/Group | 15mg MK1006/Placebo/45mg MK1006/60mg MK1006/Placebo (Fed) | Placebo/30mg MK1006/45mg MK1006/60mg MK1006/30mg MK1006 (Fed) | 15mg MK1006/30mg MK1006/Placebo/60mg MK1006/30mg MK1006 (Fed) | 15mg MK1006/30mg MK1006/45mg MK1006/Placebo/30mg MK1006 (Fed) | 60mg MK1006 / Placebo / 100mg MK1006 / 120mg MK1006 / Placebo | Placebo/80mg MK1006/100mg MK1006/120mg MK1006/140mg MK1006 | 60mg MK1006/80mg MK1006/Placebo/120mg MK1006/140mg MK1006 | 60 mg MK1006/80 mg MK1006/100 mg MK1006/Placebo/140 mg MK1006 | 140mg MK1006 / Placebo / 200mg MK1006 / 230mg MK1006 / Placebo | Placebo/170mg MK1006/200mg MK1006/230mg MK1006/260mg MK1006 | 140mg MK1006/170mg MK1006/Placebo/230mg MK1006/260mg MK1006 | 140mg MK1006/170mg MK1006/200mg MK1006/Placebo/260mg MK1006
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | 15mg MK1006/Placebo/45mg MK1006/60mg MK1006/Placebo (Fed) | Placebo/30mg MK1006/45mg MK1006/60mg MK1006/30mg MK1006 (Fed) | 15mg MK1006/30mg MK1006/Placebo/60mg MK1006/30mg MK1006 (Fed) | 15mg MK1006/30mg MK1006/45mg MK1006/Placebo/30mg MK1006 (Fed) | 60mg MK1006 / Placebo / 100mg MK1006 / 120mg MK1006 / Placebo | Placebo/80mg MK1006/100mg MK1006/120mg MK1006/140mg MK1006 | 60mg MK1006/80mg MK1006/Placebo/120mg MK1006/140mg MK1006 | 60 mg MK1006/80 mg MK1006/100 mg MK1006/Placebo/140 mg MK1006 | 140mg MK1006 / Placebo / 200mg MK1006 / 230mg MK1006 / Placebo | Placebo/170mg MK1006/200mg MK1006/230mg MK1006/260mg MK1006 | 140mg MK1006/170mg MK1006/Placebo/230mg MK1006/260mg MK1006 | 140mg MK1006/170mg MK1006/200mg MK1006/Placebo/260mg MK1006
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 (One participant discontinued after receiving the 230 mg dose of MK1006 and was not replaced) | 2 | 1 (Replacement participant discontinued after receiving placebo to 230mg MK1006 and was not replaced)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Period: Period 5
Arm/Group | 15mg MK1006/Placebo/45mg MK1006/60mg MK1006/Placebo (Fed) | Placebo/30mg MK1006/45mg MK1006/60mg MK1006/30mg MK1006 (Fed) | 15mg MK1006/30mg MK1006/Placebo/60mg MK1006/30mg MK1006 (Fed) | 15mg MK1006/30mg MK1006/45mg MK1006/Placebo/30mg MK1006 (Fed) | 60mg MK1006 / Placebo / 100mg MK1006 / 120mg MK1006 / Placebo | Placebo/80mg MK1006/100mg MK1006/120mg MK1006/140mg MK1006 | 60mg MK1006/80mg MK1006/Placebo/120mg MK1006/140mg MK1006 | 60 mg MK1006/80 mg MK1006/100 mg MK1006/Placebo/140 mg MK1006 | 140mg MK1006 / Placebo / 200mg MK1006 / 230mg MK1006 / Placebo | Placebo/170mg MK1006/200mg MK1006/230mg MK1006/260mg MK1006 | 140mg MK1006/170mg MK1006/Placebo/230mg MK1006/260mg MK1006 | 140mg MK1006/170mg MK1006/200mg MK1006/Placebo/260mg MK1006
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 1
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants were treated with MK1006 or dose-matched placebo over 5 treatment periods.
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) On Study
Description: An adverse event was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the treatment, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the treatment, was also considered an adverse experience.
Time Frame: From the time of the run-in period prior to the first dose of study drug through the end of the poststudy period (up to 3 weeks)
Population: All Participants as Treated (APaT) Population; All participants who received at least one dose of the investigational drug.
Measure: Number; unit: participants
Groups:
- 15 mg MK1006: After a minimum washout period of 7 days, participants received a single dose of 15 mg MK1006 after an overnight fast.
- 30 mg MK1006: After a minimum washout period of 7 days, participants received a single dose of 30 mg MK1006 after an overnight fast
- 45 mg MK1006: After a minimum washout period of 7 days, participants received a single dose of 45 mg MK1006 after an overnight fast.
- 60 mg MK1006: After a minimum washout period of 7 days, participants received a single dose of 60 mg MK1006 after an overnight fast.
- 80 mg MK1006: After a minimum washout period of 7 days, participants received a single dose of 80 mg MK1006 after an overnight fast.
- 100 mg MK1006: After a minimum washout period of 7 days, participants received a single dose of 100 mg MK1006 after an overnight fast.
- 120 mg MK1006: After a minimum washout period of 7 days, participants received a single dose of 120 mg MK1006 after an overnight fast.
- 140 mg MK1006: After a minimum washout period of 7 days, participants received a single dose of 140 mg MK1006 after an overnight fast.
- 170 mg MK1006: After a minimum washout period of 7 days, participants received a single dose of 170 mg MK1006 after an overnight fast.
- 200 mg MK1006: After a minimum washout period of 7 days, participants received a single dose of 200 mg MK1006 after an overnight fast.
- 230 mg MK1006: After a minimum washout period of 7 days, participants received a single dose of 230 mg MK1006 after an overnight fast.
- 260 mg MK1006: After a minimum washout period of 7 days, participants received a single dose of 260 mg MK1006 after an overnight fast.
- 30 mg MK1006 [Fed State]: After a minimum washout period of 7 days, participants received a single dose of 30 mg MK1006 after a light breakfast.
- Placebo: After a minimum washout period of 7 days, participants received a single dose of dose-matched placebo to MK1006.
Arm/Group | 15 mg MK1006 | 30 mg MK1006 | 45 mg MK1006 | 60 mg MK1006 | 80 mg MK1006 | 100 mg MK1006 | 120 mg MK1006 | 140 mg MK1006 | 170 mg MK1006 | 200 mg MK1006 | 230 mg MK1006 | 260 mg MK1006 | 30 mg MK1006 [Fed State] | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 4 | 6 | 24
participants | 2 | 3 | 3 | 2 | 2 | 1 | 1 | 5 | 1 | 3 | 2 | 3 | 2 | 13

2. Secondary Outcome: Mean Area Under the Plasma Concentration Curve From Time Zero to Infinity (AUC[0-∞]) After Single Dose MK1006
Description: The AUC(0-∞) was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity.
Time Frame: From pre-dose to 168 hours post-dose
Population: Per-Protocol (PP) Population; The subset of participants who complied with the protocol sufficiently to ensure that data was likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance included exposure to treatment, availability of measurements and absence of major protocol violations.
Measure: Mean (Standard Deviation); unit: nM.hr
Arm/Group | 15 mg MK1006 | 30 mg MK1006 | 45 mg MK1006 | 60 mg MK1006 | 80 mg MK1006 | 100 mg MK1006 | 120 mg MK1006 | 140 mg MK1006 | 170 mg MK1006 | 200 mg MK1006 | 230 mg MK1006 | 260 mg MK1006 | 30 mg MK1006 [Fed State]
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 5 | 5 | 7 | 6 | 5 | 6 | 4 | 6
nM.hr | 595 (106) | 1330 (193) | 1900 (464) | 2790 (810) | 4380 (1960) | 6360 (2680) | 7670 (1900) | 7500 (2800) | 8160 (3570) | 8440 (5520) | 11670 (4020) | 11460 (5340) | 1380 (271)
Statistical Analysis 1: Comparison: 30 mg MK1006 vs 30 mg MK1006 [Fed State]; A linear mixed-effect model was used to estimate the geometric mean AUC (0-∞) for MK1006 at every dose level; Test type: Non-Inferiority or Equivalence — To assess the effect of food at the 30 mg dose, a point estimate was constructed for the geometric mean ratio for the fed/fasted states (GMR[fed/fasted]) of MK1006 AUC (0-∞). The GMR (fed/fasted) was calculated using the geometric mean AUC (0-∞) of the fed state divided by the geometric mean AUC (0-∞) fasted state. A GMR (fed/fasted) point estimate value within 20% of unity (1.00) was considered consistent with an absence of a clinically significant food effect; Mixed-Effect Model; Geometric Mean Ratio (fed/fasted) = 1.03

3. Secondary Outcome: Mean Maximum Plasma Concentration (Cmax) of MK1006 After Single Dose
Time Frame: From pre-dose to 168 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | 15 mg MK1006 | 30 mg MK1006 | 45 mg MK1006 | 60 mg MK1006 | 80 mg MK1006 | 100 mg MK1006 | 120 mg MK1006 | 140 mg MK1006 | 170 mg MK1006 | 200 mg MK1006 | 230 mg MK1006 | 260 mg MK1006 | 30 mg MK1006 [Fed State]
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 5 | 5 | 7 | 6 | 5 | 6 | 4 | 6
nM | 60.0 (22.7) | 123.0 (27.7) | 191.0 (76.5) | 251.0 (73.4) | 434.0 (196.0) | 614.0 (267.0) | 783.0 (230.0) | 786.0 (422.) | 768.0 (364.0) | 738.0 (688.0) | 1174.0 (822.0) | 901.0 (508.0) | 141.0 (37.4)
Statistical Analysis 1: Comparison: 30 mg MK1006 vs 30 mg MK1006 [Fed State]; A linear mixed-effect model was used to estimate the geometric mean Cmax for MK1006 at every dose level; Test type: Non-Inferiority or Equivalence — To assess the effect of food at the 30 mg dose, a point estimate was constructed for the geometric mean ratio for the fed/fasted states (GMR[fed/fasted]) of MK1006 Cmax. The GMR (fed/fasted) was calculated using the geometric mean Cmax of the fed state divided by the geometric mean Cmax fasted state. A GMR (fed/fasted) point estimate value within 20% of unity (1.00) was considered consistent with an absence of a clinically significant food effect; Mixed-effect Model; Geometric Mean Ratio (fed/fasted) = 1.14

4. Secondary Outcome: Median Time of Maximum Plasma Concentration (Tmax) of MK1006 After Single Dose
Time Frame: From pre-dose to 168 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | 15 mg MK1006 | 30 mg MK1006 | 45 mg MK1006 | 60 mg MK1006 | 80 mg MK1006 | 100 mg MK1006 | 120 mg MK1006 | 140 mg MK1006 | 170 mg MK1006 | 200 mg MK1006 | 230 mg MK1006 | 260 mg MK1006 | 30 mg MK1006 [Fed State]
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 5 | 5 | 7 | 6 | 5 | 6 | 4 | 6
hr | 1.5 [1.0 to 6.0] | 2.0 [1.0 to 5.0] | 3.0 [2.0 to 5.0] | 3.0 [3.0 to 5.0] | 3.0 [2.0 to 5.0] | 3.0 [2.0 to 5.0] | 4.0 [1.0 to 5.0] | 3.0 [2.0 to 5.0] | 3.5 [1.0 to 5.0] | 5.0 [2.0 to 5.0] | 4.0 [2.0 to 5.0] | 4.5 [4.0 to 5.0] | 2.0 [2.0 to 4.0]

5. Secondary Outcome: Apparent Terminal Half-Life (T 1/2) of MK1006 After Single Dose
Description: The apparent terminal half-life was defined as the time required for the plasma concentration of MK1006 to decrease 50% in the final stage of its elimination
Time Frame: From pre-dose to 168 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | 15 mg MK1006 | 30 mg MK1006 | 45 mg MK1006 | 60 mg MK1006 | 80 mg MK1006 | 100 mg MK1006 | 120 mg MK1006 | 140 mg MK1006 | 170 mg MK1006 | 200 mg MK1006 | 230 mg MK1006 | 260 mg MK1006 | 30 mg MK1006 [Fed State]
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 5 | 5 | 7 | 6 | 5 | 6 | 4 | 6
hr | 17.0 (3.1) | 17.3 (1.3) | 17.6 (3.5) | 18.3 (2.3) | 20.0 (1.4) | 23.0 (5.2) | 19.3 (4.7) | 25.7 (5.6) | 22.3 (5.6) | 22.8 (5.0) | 26.7 (2.6) | 31.3 (6.6) | 19.2 (3.2)

6. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an AE
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 15 mg MK1006 | 30 mg MK1006 | 45 mg MK1006 | 60 mg MK1006 | 80 mg MK1006 | 100 mg MK1006 | 120 mg MK1006 | 140 mg MK1006 | 170 mg MK1006 | 200 mg MK1006 | 230 mg MK1006 | 260 mg MK1006 | 30 mg MK1006 [Fed State] | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 4 | 6 | 24
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Mean Area Under The Plasma Concentration Curve From Time Zero to 24 Hours (AUC[0-24]) After Single Dose MK1006
Description: The AUC(0-24) was estimated by determining the total area under the curve of the concentration versus time curve to 24 hours post dose.
Time Frame: From pre-dose to 168 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nM.hr
Arm/Group | 15 mg MK1006 | 30 mg MK1006 | 45 mg MK1006 | 60 mg MK1006 | 80 mg MK1006 | 100 mg MK1006 | 120 mg MK1006 | 140 mg MK1006 | 170 mg MK1006 | 200 mg MK1006 | 230 mg MK1006 | 260 mg MK1006 | 30 mg MK1006 [Fed State]
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 5 | 5 | 7 | 6 | 5 | 6 | 4 | 6
nM.hr | 468 (101) | 1030 (155) | 1520 (416) | 2100 (580) | 3450 (1570) | 4930 (2120) | 6110 (1420) | 5690 (2490) | 6590 (3320) | 6270 (4850) | 8810 (3780) | 8500 (4380) | 1060 (232)

ADVERSE EVENTS:
Time Frame: From the time of the run-in period prior to the first dose of study drug through the end of the poststudy period (up to 3 weeks)
Arm/Group | 15 mg MK1006 | 30 mg MK1006 | 45 mg MK1006 | 60 mg MK1006 | 80 mg MK1006 | 100 mg MK1006 | 120 mg MK1006 | 140 mg MK1006 | 170 mg MK1006 | 200 mg MK1006 | 230 mg MK1006 | 260 mg MK1006 | 30 mg MK1006 [Fed State] | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/4 | 0/6 | 0/24
Other Adverse Events (participants affected / at risk) | 2/6 | 3/6 | 3/6 | 2/12 | 2/6 | 1/6 | 1/6 | 5/12 | 1/6 | 3/6 | 2/6 | 3/4 | 2/6 | 12/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 15 mg MK1006 (N=6) | 30 mg MK1006 (N=6) | 45 mg MK1006 (N=6) | 60 mg MK1006 (N=12) | 80 mg MK1006 (N=6) | 100 mg MK1006 (N=6) | 120 mg MK1006 (N=6) | 140 mg MK1006 (N=12) | 170 mg MK1006 (N=6) | 200 mg MK1006 (N=6) | 230 mg MK1006 (N=6) | 260 mg MK1006 (N=4) | 30 mg MK1006 [Fed State] (N=6) | Placebo (N=24)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo Positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctival Hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry Eye (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye Pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pterygium (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Feeling Hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion Site Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis Externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
C-Reactive Protein Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T Wave Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 4
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ingrown Hair (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.